CLINICAL TRIAL: NCT00426114
Title: Acute Haemodynamic Impact of an IV Glucose-injection
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: never started due to logistic issues
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2007/016
Record Dates: First submitted 2007-01-23; First posted 2007-01-24 (Estimated); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Peritoneal Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Administration of an IV glucose-injection

SUMMARY:
Patients with peritoneal dialysis will be administered an IV glucose-injection to evaluate the haemodynamic impact of this injection. The patients will be matched with healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* Stable clinical condition
* Either peritoneal dialysis (at least one month) either matched healthy subject

Exclusion Criteria:

* Heart Failure
* Diabetes requiring insulin treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Haemodynamic parameters
Glycemia

CONTACTS AND LOCATIONS:
Overall Officials: Wim Van Biesen, MD, PhD, Principal Investigator — University Hospital, Ghent

REFERENCES:
- See also: Website of the University Hospital Ghent — http://www.uzgent.be